CLINICAL TRIAL: NCT03160378
Title: Organizational Skills Training for Children With ADHD
Acronym: OST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Region Syddanmark (Other)
Responsible Party: Principal Investigator, Aida Bikic, Ph.D., clinical psychologist, Region Syddanmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 55772 S-20160180
Record Dates: First submitted 2017-05-16; First posted 2017-05-19 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The participants in the intervention group will receive treatment as usual + 10 sessions of organizational skills training
  Interventions: Behavioral: Organizational skills training; Other: Treatment as usual
- Control (Other): Control participants will receive treatment as usual.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Organizational skills training — 10 sessions of parent and child training in a group format.
  Arms: Intervention
Other: Treatment as usual — Treatment as usual in the outpatient clinic

SUMMARY:
The purpose of this trial is to investigate the effect of organizational skills training, a parent and child training approach on organizational skills, inattentive symptoms and functional outcome in children age 6-13 years. Half of the participants will receive treatment as usual (TAU) and organizational skills training and the other half will receive TAU.

DETAILED DESCRIPTION:
Organizational skills training (OST) is a behavioral intervention that has been increasingly used to address difficulties with time management and organization of materials in children with ADHD, that tend to persist despite medication and behavioral treatments. This randomized clinical superiority trial is going to investigate the effect of Organizational Skills Training, a group treatment approach for parents and children. The program is also involving a computerized program, vTime, that will help the children manage time more effectively. A total of 98 children with ADHD aged 6-13 years is expected to be randomized to either intervention or control group in a single blind design. Both groups will receive treatment-as-usual. The intervention group is going to participate in a group training for parents and children for 10 weekly sessions.

ELIGIBILITY:
Inclusion Criteria:

1. ADHD diagnosis after clinical interview K-SADS
2. age between 6-13 years, both inclusive; informed consent.
3. The child has to score at least one standard deviation (SD) above the mean on the Plan/Organize subscale on the Behavior Rating Inventory of Executive Functions (BRIEF) (parent edition) verifying problems with organizational skills.

Exclusion Criteria:

1. autism spectrum disorder
2. serious psychopathology requiring immediate clinical attention (e.g., severe depression or aggressive behavior)
3. head injury or verified neurological disease
4. intelligence quotient (IQ <80)
5. medical condition, requiring primary treatment
6. no informed consent from custody.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 142 (Estimated)
Dates: Start 2017-05-22 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Children Organizational Skills Scale (COSS)-parent | after 10 weeks of intervention
  organizational skills questionnaire

SECONDARY OUTCOMES:
Children Organizational Skills Scale (COSS)-teacher | after 10 weeks of intervention
  organizational skills questionnaire
ADHD-Rating Scale (ADHD-RS) (parent edition) | after 10 weeks of intervention
  ADHD symptoms questionnaire
Behavior Rating Inventory of Executive Functions (BRIEF)-parent | after 10 weeks of intervention
  executive functions questionnaire
CANTAB Rapid Visual Movement (RVP) | after 10 weeks of intervention
  cognitive test
Weis's scale of disability-Parent Report (WFIRS-P) | after 10 weeks of intervention
  functional outcome questionnaire

OTHER OUTCOMES:
Behavior Rating Inventory of Executive Functions (BRIEF)-teacher | after 10 weeks of intervention
  executive functions questionnaire
CANTAB Stop Signal Task (SST) | after 10 weeks of intervention
  cognitive test
CANTAB one touch Stockings of Cambridge (SOC) | after 10 weeks of intervention
  cognitive test
CANTAB Working Memory (WM) | after 10 weeks of intervention
  cognitive test
Non-serious adverse events | after 10 weeks of intervention
  adverse events
Serious adverse events | after 10 weeks of intervention
  adverse events
Children Organizational Skills Scale (COSS)-parent | 24 weeks after ended intervention
  organizational skills questionnaire
Children Organizational Skills Scale (COSS)-teacher | 24 weeks after ended intervention
  organizational skills questionnaire
ADHD-Rating Scale (ADHD-RS) (parent edition) | 24 weeks after ended intervention
  ADHD symptoms questionnaire
ADHD-Rating Scale (ADHD-RS) (teacher edition) | 24 weeks after ended intervention
  ADHD symptoms questionnaire
Behavior Rating Inventory of Executive Functions (BRIEF)-parent | 24 weeks after ended intervention
  executive functions questionnaire
Behavior Rating Inventory of Executive Functions (BRIEF)-teacher | 24 weeks after ended intervention
  executive functions questionnaire
CANTAB Stop Signal Task (SST) | 24 weeks after ended intervention
  cognitive test
CANTAB one touch Stockings of Cambridge (SOC) | 24 weeks after ended intervention
  cognitive test
CANTAB Rapid Visual Movement (RVP) | 24 weeks after ended intervention
  cognitive test
CANTAB Working Memory (WM) | 24 weeks after ended intervention
  cognitive test
Weis's scale of disability-Parent Report (WFIRS-P) | 24 weeks after ended intervention
  functional outcome questionnaire
Non-serious adverse events | 24 weeks after ended intervention
  adverse events
Serious adverse events | 24 weeks after ended intervention
  adverse events
CANTAB Reaction time task (RTI) | after 10 weeks of intervention
  reaction time
CANTAB Reaction time task (RTI) | after 24 weeks of intervention
  reaction time
ADHD-Rating Scale (ADHD-RS) (teacher edition) | after 10 weeks of intervention
  ADHD symptoms questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Aida Bikic, Ph.D., Principal Investigator — Region of Southern Denmark and University of Southern Denmark
Locations (2):
- Denmark (2):
  - Department of Child and Adolescent Mental Health Services, Aabenraa
  - Department of Child and Adolescent Mental Health Services, Vejle

IPD SHARING:
Plan to Share IPD: Undecided
After the competition of the study, data will be stored in Danish National Archives, where data can be accessed after previous approval.

REFERENCES:
- [Derived] Bikic A, Dalsgaard S, Olsen KD, Sukhodolsky DG. Organizational skills training for children with ADHD: study protocol for a randomized, controlled trial. Trials. 2021 Oct 29;22(1):752. doi: 10.1186/s13063-021-05499-9. PMID 34715906